CLINICAL TRIAL: NCT02587143
Title: Ethyl Chloride Vapocoolant as Anesthesia for Arterial Punctures: A Randomized Clinical Trial
Brief Title: Ethyl Chloride Vapocoolant as Anesthesia for Arterial Punctures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionorte (Other)
Collaborators: Osakidetza (Other); University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, SENDOA BALLESTEROS-PEÑA, Emergency nurse practitioner, PhD doctor., Bionorte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GASOHUB
Record Dates: First submitted 2015-10-09; First posted 2015-10-27 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia; Pain
MeSH Terms: conditions — Pain | interventions — Ethyl Chloride; Methods; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Alcohol -based spray as placebo will be administrated before arterial puncture.
  Interventions: Drug: Alcohol
- Ethyl chloride (Experimental): Ethyl choride will be administrated before arterial puncture.
  Interventions: Drug: Ethyl chloride

INTERVENTIONS:
Drug: Ethyl chloride — Nurses will administrate ethyl chloride vapocoolant spray on patient's skin a few seconds before arterial puncture (of cubital arteria).
  Other Names: Intervention
  Arms: Ethyl chloride
Drug: Alcohol — Nurses will use an alcohol-based spray as placebo on patient's skin a few seconds before arterial puncture (of cubital arteria).
  Other Names: Placebo
  Arms: Control

SUMMARY:
Ethyl chloride vapocoolant sprays provide transient skin anesthesia within seconds of application. The current investigation aim is to compare the effect of ethyl chloride based vapocoolant spray to placebo in reducing pain associated with arterial puncture for gasometry determinations.

The investigators will conduce a double-blind randomized placebo-controlled trial at Emergency Department.

We will enroll patients who come to Emergency Department who need an arterial gasometry determination. Patients will be randomized to intervention-group (ethyl chloride vapocoolant sprays will be usad before arterial puncture) or to placebo-group (alcohol spray as placebo will be used before arterial puncture.) and after the puncture they will rate their pain using a 10 points visual analogue scale.

DETAILED DESCRIPTION:
Single-blind, randomized placebo-controlled trial in an emergency department of Hospital de Basurto in Bilbao, Spain. Patients for whom arterial blood gas analysis had been ordered will be included. They will be randomly assigned to receive application of the experimental ethyl chloride spray or a placebo aerosol spray of a solution of alcohol in water. The assigned spray will be applied just before arterial puncture. The main outcome variable is pain intensity reported on an 11-point numeric rating scale.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-85 years old.
* arterial gasometry determination needed
* III, IV or V level classification on Manchester triage.

Exclusion criteria:

* refusal to participate,
* inability to provide informed consent (non-Spanish speaking, dementia or altered mental state),
* skin disease associated with cold intolerance (Raynaud's phenomenon),
* known allergy to spray contents,
* Glasgow Coma Scale <15,
* pregnancy,
* under effects of alcohol or drugs,
* Allen test +.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SENDOA BALLESTEROS-PEÑA, PhD, Principal Investigator — HOSPITAL OF BASURTO (BILBAO)
Locations (1):
- Hospital de Basurto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ballesteros-Pena S, Fernandez-Aedo I, Vallejo-De la Hoz G; en representacion del Grupo de Trabajo DIASURE. [Ethyl chloride aerosol spray for local anesthesia before arterial puncture: randomized placebo-controlled trial]. Emergencias. 2017 Jun;29(3):161-166. Spanish. PMID 28825235

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seccondary effcts happens after punctre (dizziness...)
Groups:
- Ethyl Chloride: Ethyl choride will be administrated before arterial puncture.
  Ethyl chloride: Nurses will administrate ethyl chloride vapocoolant spray on patient's skin a few seconds before arterial puncture.
- Control: Alcohol -based spray as placebo will be administrated before arterial puncture.
  Alcohol: Nurses will use an alcohol-based spray as placebo on patient's skin a few seconds before arterial puncture.
Period: Overall Study
Arm/Group | Ethyl Chloride | Control
Started | 66 | 60
Completed | 65 | 60
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ethyl Chloride | Total
Number analyzed (Participants) | 60 | 66 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (12.1) | 67.1 (14.4) | 67.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 38 | 41 | 79
Arteria of puncture [Count of Participants; unit: Participants] — Puncture on humeral arteria or cubital arteria
  Participants
    Cubital arteria | 50 | 56 | 106
    Humeral arteria | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Level on the Visual Analog Scale (NRS-11)
Description: patients will measure their pain score on a visual analog scale (NRS-11: Numeric Rate Score, from 0 -no pain- to 10 points -the worst pain ever-) after the puncture
Time Frame: scores on a scale immediately after the puncture
Measure: Median (Inter-Quartile Range); unit: scores on scale
Arm/Group | Control | Ethyl Chloride
Number analyzed (Participants) | 60 | 66
scores on scale | 2 [1 to 4.5] | 2 [1 to 5]

ADVERSE EVENTS:
Arm/Group | Control | Ethyl Chloride
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/66
Other Adverse Events (participants affected / at risk) | 0/60 | 1/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=60) | Ethyl Chloride (N=66)
Local injury (ischaemia) (Vascular disorders) | 0 (0) | 0 (0)
Dizziness after puncture (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No